CLINICAL TRIAL: NCT00811967
Title: Inhibition of Disease Progression in Hepatitis C-infected Patients With Compensated Liver Cirrhosis
Brief Title: Inhibition of Disease Progression in Hepatitis C-infected Patients With Compensated Liver Cirrhosis (P03811) (COMPLETED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03811; JPC-02-320-34
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental)
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)
- Control Arm (No Intervention)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron administered at a dose of 1.5 ug/kg QW SC for up to 48 weeks
  Other Names: SCH 54031
  Arms: Treatment Arm
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered at a dose of 600, 800, or 1000 mg/day, orally, for up to 48 weeks.
  Other Names: SCH 18908
  Arms: Treatment Arm

SUMMARY:
The objective of the study is to evaluate the superiority of treatment with PegIntron and Rebetol over no antiviral therapy (control group) in subjects with chronic hepatitis C and type C compensated cirrhosis. Subjects will be randomized in a ratio of 2:1 (Treatment Arm to Control Arm). Subjects in the Treatment Arm will receive combination therapy with PegIntron and Rebetol for 48 weeks; then will enter a 24-week post-treatment Follow-up. Subjects who have detectable Hepatitis C Virus-RNA at Treatment Week 24 will discontinue treatment and enter Follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with compensated hepatic cirrhosis secondary to chronic hepatitis C who would meet all the inclusion criteria below and would not interfere with any of the exclusion criteria below.

* Patients (regardless of gender) who can take contraceptive measures from date of informed consent to the end of follow-up
* Patients who meet all the criteria below in the test/observation/ investigation in 30 days before the beginning of treatment.

  * Patients with quantitative HCV-RNA (+)
  * ALT > 40 IU/L
  * Patients who are classified as Child-Pugh Classification A, and who do not have ascites or hepatic encephalopathy
  * Prothrombin Time <=3.0 seconds prolonged, total bilirubin <= 1.5 mg/dL or direct bilirubin <= 0.7 mg/dL, Albumin >= 3.0 g/dL
  * AFP within normal limits, AFP-L3 <= 10%，PIVKA-II <= 100 mAU/mL
  * Serum creatinine <= upper limit of normal, creatinine clearance >= 51 mL/minute
  * Patients with fasting blood glucose < 110 mg/dL.
  * Thyroid-stimulating hormone within normal limits
  * Hemoglobin level >= 12 g/dL，leukocyte count >= 3,000/mm3，neutrophil count >= 1,500 /mm3，platelet count >= 80,000/mm3
* Patients who weighs more than 40 kg and not more than 100 kg within 60 days prior to registration
* Patients who were diagnosed with liver cirrhosis (fibrosis score: F4) based on the liver biopsy performed within a year prior to registration and is able to provide with liver tissue sample.
* Patients who between the ages of 20 and 70 years at time of informed consent who can give written informed consent
* Patients who can be hospitalized at least for 14 days from the initiation of treatment.

Exclusion Criteria:

* Patients who have been administered pegylated interferon or ribavirin in the past.
* Patients who had previously received treatment with IFN for whom at least 90 days have not elapsed since the end of previous treatment by the time of registration in the study
* Patients who have received treatment within 14 days prior to registration with the injectable preparations containing glycyrrhizin/cysteine/glycyron (Stronger Neo-Minophagen C, etc.), or shosaikoto
* Patients who have had antiviral drug or antitumor drug, or immune regulation therapy (including steroid administration, radiation therapy) within 90 days prior to registration. [except for topical application and external drug]
* Patients who have been administered any study drug within 180 days prior to registration.
* Patients who meet the following criteria in the screening test

  * HBs antigen positive
  * antinuclear antibody >= 320 times
* Patients with or who have a history of primary biliary cirrhosis, hepatic failure, hepatocellular carcinoma.
* Patients with other etiologies of liver disease such as autoimmune, alcoholic and drug-induced liver diseases
* Patients with or who have a history of decompensated cirrhosis with following disorder. Ascites, jaundice, bleeding varices, esophageal and/or gastric varices which needs treatment, hepatic encephalopathy, and spontaneous bacterial peritonitis.
* Patients with hemophilia
* Patients with or who have a history of neuropsychiatry disorder such as depression.
* Patients with or who have a history of epileptic seizures requiring treatment
* Patients with or who have a history of angina pectoris, heart failure, myocardial infarction, uncontrollable hypertension (diastolic blood pressure: equal to or more than 110mmHg) or arrhythmia which needs treatment.
* Patients with chronic pulmonary disease
* Patients with or who have a history of autoimmune disease (Crohn's disease, ulcerative colitis, chronic rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, etc).
* Patients with Hemoglobinopathies (thalassaemia, sickle cell anemia)
* Patients with malignant tumors
* Patients with organ transplants (other than cornea and hair transplant).
* Patients with a history of hypersensitivity to interferon preparations, biological products such as vaccine, or nucleoside analogs
* Female patients who are pregnant or nursing (male patients with partner who are pregnant), and for whom pregnancy cannot be ruled out by serum HCG test conducted during the screening period
* Patients with specific reaction to PEG-IFNα-2b in prick test conducted before the initiation of treatment（Only PEG/R group）
* Other patients judged by the investigator (sub-investigator) to be inappropriate for inclusion in this study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response rate, defined as the proportion of subjects with undetectable HCV-RNA at 24-week post-treatment follow-up | Measured at 24 weeks post-treatment

SECONDARY OUTCOMES:
Rate of subject with undetectable HCV-RNA at the end of treatment (or at discontinuation of treatment) | Measured at the end of treatment (or at discontinuation of treatment)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html